CLINICAL TRIAL: NCT04207541
Title: Promoting Insulin Acceptance and Initiation With the Tailor-made Educational Intervention Among Type 2 Diabetic Patients With Sub-optimal Glycemic Control
Brief Title: Promoting Insulin Initiation Among Suboptimal Diabetic Control Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Echo Ting-Ting Go, Doctoral Candidate, The University of Hong Kong
Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: UW 19-614
Record Dates: First submitted 2019-10-30; First posted 2019-12-23 (Actual); Last update posted 2019-12-23 (Actual); Status verified 2019-12

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 diabetes; insulin initiation; Brief motivational interview; Psychological insulin resistance
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Recruit control group first then interventional group.
Masking Description: Participant does not know which group they are assigned to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Control group and Intervention group (Experimental): For control group, participants will be treated with usual care. For intervention group, participants will be provided a session of education regarding insulin initiation with brief motivation interviewing.
  Interventions: Behavioral: Brief motivational interview

INTERVENTIONS:
Behavioral: Brief motivational interview — Client (who has suboptimal diabetic control with oral anti-diabetic agent) will be advised for insulin initiation with brief motivational interviewing in one session of individual education.

SUMMARY:
Delay in commencing insulin among type 2 Diabetes Mellitus (T2DM) patients is common. One of the reasons is patients' psychological insulin resistance (PIR), which is particularly prevalent in Chinese patients. The Chinese Attitudes to Starting Insulin Questionnaire (Ch-ASIQ) is the shortest locally validated questionnaire which is developed to understand the condition of PIR in T2DM patients while brief motivational interviewing has been shown to improve patients' collaborations and satisfactions, the alliance between patients and doctors, and the treatment adherence. Therefore, this study aims to investigate the efficacy of a one-session educational intervention targeting psychological insulin resistance guided by Ch-ASIQ in promoting the insulin acceptance and initiation.

A quasi-experimental study will be conducted on 130 insulin-naïve T2DM patients recruited from a primary care setting. Eligible participants in the intervention group will be treated with one 15-minute brief motivational interviewing guided by Ch-ASIQ while those in control group will be treated with usual care. Both groups will be further followed up for 6 months to observe for their insulin initiation. The primary outcomes: i. the proportion of patient referral to insulin clinic (insulin acceptance), and ii. the proportion of patient with insulin initiation (actual start of insulin therapy).

DETAILED DESCRIPTION:
Background Information According to the American Diabetes Association ADA (2018), insulin treatment should not be delayed in patients with T2DM who fail to control their glycemic level with OHAs. Delay in insulin therapy for such type of patients leads to excess glycemic burden. A retrospective analysis of data showed that between 2005 and 2010, the time from T2DM diagnosis to insulin initiation increased by approximately 2 years in the primary care practices in Europe with increase in the percentage of patients with at least one macrovascular complication. As known, once the developed macrovascular complications cannot be reversed with tight glycemic control by any treatment. However, the initiation of the insulin therapy is often delayed. This may be due to the reluctance among people with T2DM.

About half of the diabetic patients who are having suboptimal glycemic control for 3-5 years and living with different extent of complications delay insulin therapy initiation. One of the reasons is patients' psychological insulin resistance (PIR), which is describing the reluctance to initiate insulin therapy, particularly prevalent in Chinese patients. In Hong Kong, a local study has revealed a similarly high PIR prevalence of 72.1%.

Effective educational programmes are needed for insulin-naive patients to enhance their understanding of the disease and treatment; and increase the acceptance and adherence of insulin therapy. This calls for effective educational programmes to help those patients in achieving better glycemic control in order to decrease risk of diabetic complications.

Brief Motivational Interviewing is an adaptation of motivational interviewing skills, which is designed to apply in a time-constraint clinical care environment and has been shown to improve patients' collaborations and satisfactions, the alliance between patients and doctors, and the adherence to treatment. Although this is an effective communication style, it has never been applied to educational programmes of insulin acceptance among T2DM patients with sub-optimal glycemic control.

Trial Objectives and Purpose This trial is to examine the effectiveness of brief motivational enhancement education programme in addition to usual care versus usual care only in improving insulin acceptance and insulin initiation among T2DM patients with sub-optimal glycemic control.

Trial Design To achieve the objectives, a quasi-experimental study on brief motivational enhancement education programme will be conducted.

Selection and Withdrawal of Subjects

Subjects will be included in the trial if they are:

1. Diagnosed with T2DM for more than six months
2. Chinese patients who can speak Cantonese/Mandarin
3. Chinese patients who can read Chinese
4. Aged ≥ 18 years
5. Suboptimal glycemic control whose latest HbA1c ≥ 7.5% with maximum oral dosage of OHAs.
6. Never used insulin before and prescribed to start insulin therapy

People will be excluded if they are:

1. Physical or mental ill that hindered them from completing the questionnaire or communicate, e.g., dementia, deafness, and severe visual problems
2. Pregnant
3. Gestational diabetic patients

People has the right to withdraw from the trial at any time without any impact on the current medical services and legal rights.

The study will be conducted in one of the primary care setting of Hospital Authority, Ap Lei Chau GOPC. Potential participants will be invited to participate when they are attending the clinic for their regular follow-up appointment. Eligible participants will first be explained the information sheet regarding the study. They will then be asked to sign the consent if they are willing to join the study.

Treatment of Subjects The study target to recruit two groups of eligible cases. The two groups will be recruited one by one. The first group recruited will act as control in comparison. In this group, all eligible participants will be invited to complete the 13-items Chinese Attitudes to Starting Insulin Questionnaire (Ch-ASIQ) before they see nurses. After having completed the questionnaires, they will be treated as usual care. The complications of suboptimal diabetic control will be told, at the same time, diet control and importance of regular exercise will also be reinforced as usual care. At the end of the session, they will be asked if they accept the referral to the insulin clinic for insulin therapy.

The interventional group of eligible cases will be recruited after the control group reached the pre-set numbers. In the interventional group, the eligible participants will be also invited to complete the Ch-ASIQ before they see nurses. Besides the usual care, all the participants in this group will also be treated with structured intervention. The information gathered through the questionnaires will be used in the intervention for this group of patients. The information will be delivered to the patients in the format of one 15-minute session of brief motivational interviewing. Pre-set script will be used for the brief motivational interviewing. At the end of the session, they will be asked if they accept the referral to the insulin clinic for insulin therapy.

The first 10 cases in the intervention group will act as pilot. Intervention will be revised if there are logistics problem seen.

ELIGIBILITY:
Inclusion Criteria:

Subjects will be included in the trial if they are:

1. Diagnosed with T2DM for more than six months
2. Chinese patients who can speak Cantonese/Mandarin
3. Chinese patients who can read Chinese
4. Aged ≥ 18 years
5. Suboptimal glycemic control whose latest HbA1c ≥ 7.5% with maximum oral dosage of OHAs.
6. Never used insulin before and prescribed to start insulin therapy

Exclusion Criteria:

People will be excluded if they are:

1. Physical or mental ill that hindered them from completing the questionnaire or communicate, e.g., dementia, deafness, and severe visual problems
2. Pregnant
3. Gestational diabetic patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of insulin acceptance | The acceptance is assessed on the same day of recruitment after education session has been provided to the participants.
  It is related to the proportion of participants who agree to be referred to insulin clinic for considering insulin initiation.
Proportion of insulin initiation | For those participants who start insulin therapy in 6 months after the education session will be regarded as "insulin initiation".
  It is related to the proportion of participants who agree to start insulin therapy after attending the insulin clinic.

CONTACTS AND LOCATIONS:
Overall Officials: Echo Ting Ting Go, Nursing, Principal Investigator — The University of Hong Kong
Locations (1):
- Hospital Authority, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No